CLINICAL TRIAL: NCT02924883
Title: A Randomized, Multicenter, Double-Blind, Placebo-Controlled Phase II Study of the Efficacy and Safety of Trastuzumab Emtansine in Combination With Atezolizumab or Atezolizumab-Placebo in Patients With HER2-Positive Locally Advanced or Metastatic Breast Cancer Who Have Received Prior Trastuzumab and Taxane Based Therapy
Brief Title: A Study to Evaluate the Efficacy and Safety of Trastuzumab Emtansine in Combination With Atezolizumab or Atezolizumab-Placebo in Participants With Human Epidermal Growth Factor-2 (HER2) Positive Locally Advanced or Metastatic Breast Cancer (BC) Who Received Prior Trastuzumab and Taxane Based Therapy
Acronym: KATE2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WO30085; 2015-004189-27 (EudraCT Number)
Record Dates: First submitted 2016-09-21; First posted 2016-10-05 (Estimated); Results first posted 2019-02-12 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-01

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — atezolizumab; Ado-Trastuzumab Emtansine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Trastuzumab Emtansine + Atezolizumab (Experimental): Atezolizumab 1200 milligrams (mg) intravenous (IV) infusion or matching Placebo followed by trastuzumab emtansine 3.6 milligrams per kilogram (mg/kg) IV infusion on Day 1 Cycle 1 and thereafter on Day 1 of each 21-day cycle until disease progression, unmanageable toxicity, or study termination by the Sponsor (approximately 29 months)
  Interventions: Drug: Atezolizumab; Drug: Trastuzumab emtansine; Other: Placebo
- Trastuzumab Emtansine + Placebo (Active Comparator): Placebo matched to atezolizumab followed by trastuzumab emtansine 3.6 mg/kg IV infusion on Day 1 Cycle 1 and thereafter on Day 1 of each 21-day cycle until disease progression, unmanageable toxicity, or study termination by the sponsor (approximately 29 months)
  Interventions: Drug: Trastuzumab emtansine; Other: Placebo

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab 1200 mg IV infusion
  Other Names: Tecentriq, RO5541267, MPDL3280A
  Arms: Trastuzumab Emtansine + Atezolizumab
Drug: Trastuzumab emtansine — Trastuzumab emtansine 3.6 mg/kg IV infusion
  Other Names: Kadcyla®, T-DM1, RO5304020
Other: Placebo — Placebo matched to atezolizumab

SUMMARY:
This Phase II, double-blind, randomized, placebo-controlled multicenter study will investigate the efficacy and safety of trastuzumab emtansine in combination with atezolizumab or atezolizumab-placebo in participants with HER2-positive locally advanced or metastatic BC who have received prior trastuzumab and taxane based therapy, either alone or in combination, and/or who have progressed within 6 months after completing adjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

* Archival tumor samples must be obtained from primary and/or metastatic sites
* Able to submit tumor tissue that is evaluable for programmed death- ligand 1 (PD-L1) expression
* HER-2 positive BC as defined by an immunohistochemistry score of 3 or gene amplified by in-situ hybridization as defined by a ratio of greater than or equal to (>=) 2.0 for the number of HER2 gene copies to the number of chromosome 17 copies
* Histologically or cytologically confirmed invasive BC: incurable, unresectable, locally advanced BC previously treated with multimodality therapy or metastatic BC
* Prior treatment for BC in the: adjuvant; unresectable locally advanced; or metastatic settings; which must include both, a taxane and trastuzumab (alone or in combination with another agent)
* Progression must have occurred during or after most recent treatment for locally advanced/metastatic BC or within 6 months after completing adjuvant therapy
* Participants must have measurable disease that is evaluable as per RECIST v1.1
* Eastern Cooperative Oncology Group Performance Status of 0 or 1
* Negative serum pregnancy test within 7 days of enrollment for pre-menopausal women and for women less than 12 months after the onset of menopause
* Use of highly effective method of contraception as defined by the protocol

Exclusion Criteria:

* Prior treatment with trastuzumab emtansine, cluster of differentiation 137 agonists, anti-programmed death-1, or anti-PD-L1 therapeutic antibody or pathway-targeting agents
* Receipt of any anti-cancer drug/biologic or investigational treatment within 21 days prior to Cycle 1 Day 1 except hormone therapy, which can be given up to 7 days prior to Cycle 1 Day 1; recovery of treatment related toxicity consistent with other eligibility criteria
* Radiation therapy within 2 weeks prior to Cycle 1, Day 1
* History of exposure to the cumulative doses of anthracyclines
* History of other malignancy within the previous 5 years, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, Stage I uterine cancer, or participants who have undergone potentially curative therapy with no evidence of disease and are deemed by the treating physician to be at low risk for recurrence
* Cardiopulmonary dysfunction, symptomatic pleural effusion, pericardial effusion, or ascites
* Participants with severe infection within 4 weeks prior to randomization, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia
* Current severe, uncontrolled systemic disease
* Major surgical procedure or significant traumatic injury within 28 days prior to randomization or anticipation of the need for major surgery during the course of study treatment
* Clinically significant history of liver disease, including cirrhosis, current alcohol abuse, autoimmune hepatic disorders, sclerosis cholangitis or active infection with human immunodeficiency virus, hepatitis B virus, or hepatitis C virus
* Need for current chronic corticosteroid therapy (>=10 mg of prednisone per day or an equivalent dose of other anti-inflammatory corticosteroids)
* Spinal cord compression not definitively treated with surgery and/or radiation, or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for greater than (>) 2 weeks prior to randomization
* Participants with known central nervous system disease
* Leptomeningeal disease
* History of autoimmune disease
* Prior allogeneic stem cell or solid organ transplantation
* Active tuberculosis
* Receipt of a live, attenuated vaccine within 4 weeks prior to randomization or anticipation that such a live, attenuated vaccine will be required during the study
* Treatment with systemic immunostimulatory agents within 4 weeks or five half-lives of the drug (whichever is shorter) prior to randomization
* Treatment with systemic corticosteroids or other systemic immunosuppressive medications within 2 weeks prior to randomization, or anticipated requirement for systemic immunosuppressive medications during the trial
* Participants who are breastfeeding, or intending to become pregnant during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2016-09-26 (Actual); Primary Completion 2017-12-11 (Actual); Study Completion 2020-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (68):
- United States (15):
  - Breastlink Med Group Inc, Orange, California
  - University of Colorado, Aurora, Colorado
  - MedStar Georgetown University Hospital (Lombardi Comprehensive Cancer Center), Washington D.C., District of Columbia
  - SCRI Florida Cancer Specialists South, Fort Myers, Florida
  - Florida Cancer Specialists; Saint Petersburg, St. Petersburg, Florida
  - Northside Hospital, Atlanta, Georgia
  - Johns Hopkins Univ Med Center, Baltimore, Maryland
  - San Juan Oncology Associates, Farmington, New Mexico
  - Laura and ISAAC Perlmutter Cancer Center at NYU Langone., New York, New York
  - Ohio State Uni Medical Center, Columbus, Ohio
  - Magee Womens Hospital, Pittsburgh, Pennsylvania
  - Cancer Care Associates of York, York, Pennsylvania
  - SCRI Tennessee Oncology Chattanooga, Chattanooga, Tennessee
  - Tennessee Oncology; Sarah Cannon Research Institute, Nashville, Tennessee
  - University of Washington, Seattle, Washington
- Australia (7):
  - St George Hospital; Cancer Care Centre, Kogarah, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Princess Alexandra Hospital Woolloongabba; Clinical Hematology and Medical Oncology, Woolloongabba, Queensland
  - Peter MacCallum Cancer Center, East Melbourne, Victoria
  - Peninsula and South Eastern Haematology and Oncology Group, Frankston, Victoria
  - Sunshine Hospital, St Albans, Victoria
  - St John of God Hospital; Bendat Cancer Centre, Subiaco, Western Australia
- Canada (6):
  - Lakeridge Health Oshawa; Oncology, Oshawa, Ontario
  - The Ottawa Hospital Cancer Centre; Oncology, Ottawa, Ontario
  - Sunnybrook Odette Cancer Centre, Toronto, Ontario
  - McGill University; Sir Mortimer B Davis Jewish General Hospital; Oncology, Montreal, Quebec
  - McGill University; Glen Site; Oncology, Montreal, Quebec
  - Hopital du Saint Sacrement, Québec, Quebec
- Germany (6):
  - HELIOS Klinikum Berlin-Buch; Klinik für Gynäkologie und Geburtshilfe, Berlin
  - Studienzentrum Berlin City, Berlin
  - Klinikum Essen-Mitte Ev. Huyssens-Stiftung / Knappschafts GmbH; Klinik für Senologie / Brustzentrum, Essen
  - Praxis für Interdisziplinäre Onkologie und Hämatologie GbR, Freiburg im Breisgau
  - Nationales Centrum für Tumorerkrankungen (NCT) ; Gyn. Onk. Frauenklinik; Uniklinikum Heidelberg, Heidelberg
  - Institut für Versorgungsforschung in der Onkologie GbR Koblenz, Koblenz
- Italy (6):
  - IRCCS Istituto Nazionale Tumori Fondazione Pascale; Oncologia Medica A, Napoli, Campania
  - A.O.U Policlinico S. Orsola Malpighi di Bologna U.O di Medicina Interna Borghi - Pad.2, Bologna, Emilia-Romagna
  - Ospedale Regionale Di Parma; Divisione Di Oncologia Medica, Parma, Emilia-Romagna
  - Centro Di Riferimento Oncologico; SOC Oncologia Medica C, Aviano, Friuli Venezia Giulia
  - Centro Catanese Di Oncologia; Oncologia Medica, Catania, Sicily
  - Ospedale Santo Stefano, Azienda USL Centro Prato, Prato, Tuscany
- South Korea (5):
  - National Cancer Center, Goyang-si
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
- Spain (6):
  - Hospital Universitario Reina Sofia; Servicio de Oncologia, Córdoba, Cordoba
  - Complejo Hospitalario Universitario A Coruña (CHUAC, Materno Infantil), Oncología, A Coruña
  - Hospital Univ Vall d'Hebron; Servicio de Oncologia, Barcelona
  - Hospital Ramon y Cajal; Servicio de Oncologia, Madrid
  - Hospital Clinico Universitario de Valencia; Servicio de Onco-hematologia, Valencia
  - Hospital Arnau de Vilanova (Valencia) Servicio de Oncologia, Valencia
- Taiwan (8):
  - Changhua Christian Hospital; Dept of Surgery, Changhua
  - Kaohsiung Medical Uni Chung-Ho Hospital; Dept of Surgery, Kaohsiung City
  - China Medical University Hospital; Surgery, Taichung
  - Chi-Mei Medical Center, Tainan
  - VETERANS GENERAL HOSPITAL; Department of General Surgery, Taipei
  - National Taiwan Uni Hospital; General Surgery, Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center; Hemato-Oncology, Taipei
  - Chang Gung Memorial Hospital - Linkou, Taoyuan District
- United Kingdom (9):
  - Royal United Hospital; Oncology Department, Bath
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Royal Free Hospital; Dept of Oncology, London
  - Royal Marsden Hosp NHS Fnd; Breast Unit, London
  - Christie Hospital; Breast Cancer Research Office, Manchester
  - Nottingham City Hospital, Nottingham
  - Weston Park Hospital; Cancer Clinical Trials Centre, Sheffield
  - Royal Marsden Hosp NHS Fnd; Medicine - Breast Unit, Sutton
  - Singleton Hospital; Pharmacy, Swansea

REFERENCES:
- [Derived] Emens LA, Esteva FJ, Beresford M, Saura C, De Laurentiis M, Kim SB, Im SA, Wang Y, Salgado R, Mani A, Shah J, Lambertini C, Liu H, de Haas SL, Patre M, Loi S. Trastuzumab emtansine plus atezolizumab versus trastuzumab emtansine plus placebo in previously treated, HER2-positive advanced breast cancer (KATE2): a phase 2, multicentre, randomised, double-blind trial. Lancet Oncol. 2020 Oct;21(10):1283-1295. doi: 10.1016/S1470-2045(20)30465-4. PMID 33002436

RESULTS

PARTICIPANT FLOW:
Groups:
- Trastuzumab Emtansine + Atezolizumab: Atezolizumab 1200 milligrams (mg) intravenous (IV) infusion followed by trastuzumab emtansine 3.6 milligrams per kilogram (mg/kg) IV infusion on Day 1 Cycle 1 and thereafter on Day 1 of each 21-day cycle until disease progression, unmanageable toxicity, or study termination by the Sponsor (up to study duration of approximately 40 months)
- Trastuzumab Emtansine + Placebo: Placebo matched to atezolizumab followed by trastuzumab emtansine 3.6 mg/kg IV infusion on Day 1 Cycle 1 and thereafter on Day 1 of each 21-day cycle until disease progression, unmanageable toxicity, or study termination by the sponsor (up to study duration of approximately 40 months)
Period: Overall Study
Arm/Group | Trastuzumab Emtansine + Atezolizumab | Trastuzumab Emtansine + Placebo
Started | 133 | 69
Completed | 0 | 0
Not Completed | 133 | 69
Not completed — Death | 39 | 20
Not completed — Lost to Follow-up | 1 | 0
Not completed — Symptomatic Deterioration/ Clinical Progression | 0 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 22 | 16
Not completed — Progressive Disease | 1 | 0
Not completed — Study Terminated by Sponsor | 69 | 32

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Trastuzumab Emtansine + Atezolizumab | Trastuzumab Emtansine + Placebo | Total
Number analyzed (Participants) | 133 | 69 | 202
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.7 (9.9) | 54.4 (10.9) | 53.9 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 131 | 69 | 200
  Male | 2 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 1 | 11
  Not Hispanic or Latino | 114 | 66 | 180
  Unknown or Not Reported | 9 | 2 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 49 | 23 | 72
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 5 | 1 | 6
  White | 72 | 44 | 116
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 5 | 1 | 6
Region [Number; unit: Number of Participants]
  USA | 21 | 11 | 32
  Western Europe | 50 | 26 | 76
  Rest of the World | 62 | 32 | 94
Programmed Cell-Death Ligand 1 Immunohistochemistry status [Number; unit: Number of Participants]
  PD-L1 positive | 57 | 27 | 84
  PD-L1 negative | 76 | 42 | 118

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) as Determined by Investigator's Tumor Assessment Using Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 (v1.1)
Description: PFS was defined as the time from randomization to the first occurrence of disease progression or death from any cause, whichever occurred first, on the basis of investigator assessments. Progression was defined as at least a 20% increase in the sum of diameters of target lesions with an absolute increase of at least 5 millimeter (mm) or the appearance of one or more new lesions.
Time Frame: Baseline up to approximately 15 months
Population: The intent-to-treat (ITT) population included all randomized participants grouped according to the treatment assigned at randomization.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab Emtansine + Placebo | Trastuzumab Emtansine + Atezolizumab
Number analyzed (Participants) | 69 | 133
months | 6.8 [4.0 to 11.1] | 8.2 [5.8 to 10.7]
Statistical Analysis 1: Comparison: Trastuzumab Emtansine + Placebo vs Trastuzumab Emtansine + Atezolizumab; Test type: Superiority; p = 0.3332, Log Rank; The 2-sided log-rank test, was stratified by world region (Western Europe vs U.S. vs Rest of World) and PD-L1 status (IC 0 vs IC 1/2/3); Hazard Ratio (HR) = 0.82, 95% CI [0.55 to 1.23]

2. Primary Outcome: Percentage of Participants With Adverse Events
Description: An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time Frame: Baseline up to study completion, approximately 40 months
Population: The safety analysis population consisted of all participants who received at least one dose of study drug. Safety analyses were based on the treatment that participants actually received.
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab Emtansine + Placebo | Trastuzumab Emtansine + Atezolizumab
Number analyzed (Participants) | 68 | 132
percentage of participants | 97.0 | 99.2

3. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death from any cause.
Time Frame: Baseline up to study completion or death, whichever occurs first, approximately 40 months
Population: The ITT population included all randomized participants grouped according to the treatment assigned at randomization.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trastuzumab Emtansine + Placebo | Trastuzumab Emtansine + Atezolizumab
Number analyzed (Participants) | 69 | 133
Months | NA [NA to NA] — Median and corresponding 95% CI could not be estimated as too few patients had an event. | NA [NA to NA] — Median and corresponding 95% CI could not be estimated as too few patients had an event.
Statistical Analysis 1: Comparison: Trastuzumab Emtansine + Placebo vs Trastuzumab Emtansine + Atezolizumab; Test type: Superiority; p = 0.2934, Log Rank; The 2-sided log-rank test was stratified by world region (Western Europe vs U.S. vs Rest of World) and PD-L1 status (IC 0 vs IC 1/2/3); Hazard Ratio (HR) = 0.74, 95% CI [0.42 to 1.30]

4. Secondary Outcome: Percentage of Participants With Objective Response (OR) as Determined by Investigator's Tumor Assessment Using RECIST v1.1
Description: An OR was defined as a complete or partial response determined on 2 consecutive occasions ≥ 4 weeks apart using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Complete response was defined as the disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) must be < 10 mm on the short axis. Partial response was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum. Participants who had no post-baseline tumor assessment were counted as non-responders.
Time Frame: Baseline up to approximately 15 months
Population: The ITT population included all randomized participants grouped according to the treatment assigned at randomization. In Participants with baseline measurable disease were considered for OR. In the atezolizumab arm, one patient was not ORR evaluable.
Measure: Number; unit: Percentage of participants
Arm/Group | Trastuzumab Emtansine + Placebo | Trastuzumab Emtansine + Atezolizumab
Number analyzed (Participants) | 69 | 132
Percentage of participants | 43.5 | 45.5

5. Secondary Outcome: Duration of OR as Determined by Investigator's Tumor Assessment Using RECIST v1.1
Description: Duration of OR was defined as the time from the first tumor assessment that was judged to indicate that the patient had an objective response to the time of first documented disease progression using RECIST v1.1 per investigator assessment or death from any cause, whichever occurred first.
Time Frame: Baseline up to approximately 15 months
Population: The ITT population included all randomized participants grouped according to the treatment assigned at randomization. Participants with OR were considered for duration of OR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trastuzumab Emtansine + Placebo | Trastuzumab Emtansine + Atezolizumab
Number analyzed (Participants) | 69 | 133
Months | NA [9.9 to NA] — Median and upper bound of 95% CI could not be estimated as too few patients had an event. | NA [7.1 to NA] — Median and upper bound of 95% CI could not be estimated as too few patients had an event.
Statistical Analysis 1: Comparison: Trastuzumab Emtansine + Placebo vs Trastuzumab Emtansine + Atezolizumab; Test type: Superiority; p = 0.6099, Log Rank; Stratified Cox proportional hazards model was stratified by world region (Western Europe, U.S., Rest of World) and PD-L1 status (IC 0, IC 1/2/3); Hazard Ratio (HR) = 1.26, 95% CI [0.52 to 3.03]

6. Secondary Outcome: Maximum Serum Concentration (Cmax) of Trastuzumab Emtansine
Description: Average post infusion Trastuzumab Emtansine concentration
Time Frame: Pre-infusion (0 hour [h]), 30 minutes (min) after end of infusion (EOI) (over 90 min) on Day 1 Cycles 1 and 4; pre-infusion (0 h) on Day 1 Cycle 2 (each cycle = 21 days); at any time during study treatment/early discontinuation visit (approx. 40 months)
Population: PK population included all participants who received at least one dose of trastuzumab emtansine with at least one post-dose concentration data point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Trastuzumab Emtansine + Atezolizumab | Trastuzumab Emtansine + Placebo
Number analyzed (Participants) | 110 | 50
ug/mL | 63.9 (116.9) | 73.2 (47.5)

7. Secondary Outcome: Cmax of Deacetyl Mercapto 1-Oxopropyl Maytansine (DM1)
Description: Average post infusion Deacetyl Mercapto 1-Oxopropyl Maytansine concentration of trastuzumab emtansine infusion
Time Frame: Pre-infusion (0 h) on Day 1 Cycle 1 and 30 min after EOI (over 90 min) on Day 1 Cycles 1 and 4 (each cycle = 21 days)
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Trastuzumab Emtansine + Placebo | Trastuzumab Emtansine + Atezolizumab
Number analyzed (Participants) | 24 | 37
ng/mL | 3.19 (84.7) | 4.21 (89.5)

8. Secondary Outcome: Cmax of Total Trastuzumab
Time Frame: Pre-infusion (0 h), 30 min after EOI (over 90 min) on Day 1 Cycles 1 and 4; pre-infusion (0 h) on Day 1 Cycle 2 (each cycle = 21 days)
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Trastuzumab Emtansine + Placebo | Trastuzumab Emtansine + Atezolizumab
Number analyzed (Participants) | 50 | 110
ug/mL | 86.5 (26.4) | 79.5 (58.3)

9. Secondary Outcome: Cmax of Atezolizumab
Description: Average post infusion atezolizumab concentration
Time Frame: Pre-infusion (0 h), 30 min after EOI (over 60 min) on Day 1 Cycles 1 and 4; pre-infusion (0 h) on Day 1 Cycles 2, 3, 8, and every 8 cycles thereafter (each cycle=21 days) up to 120 days after treatment completion/early discontinuation (approx. 40 months)
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Trastuzumab Emtansine + Atezolizumab
Number analyzed (Participants) | 98
ug/mL | 626 (23.0)

10. Secondary Outcome: Percentage of Participants With Anti-therapeutic Antibodies (ATAs) to Atezolizumab
Description: ATAs are antibodies that inactivate the therapeutic effects of Atezolizumab. Patients are considered to be ATA positive if they are ATA negative at baseline but develop an ATA response following study drug administration (treatment-induced ATA response), or if they are ATA positive at baseline and the titer of one or more post-baseline samples is at least 4-fold greater (i.e., ≥ 0.60 titer units) than the titer of the baseline sample (treatment-enhanced ATA response).
Time Frame: Pre-infusion (0 h) on Day 1 Cycles 1, 2, 3, 4, 8, and every 8 cycles thereafter (each cycle = 21 days) up to 120 days after treatment completion or early discontinuation (approximately 40 months)
Population: The analysis population included a patient with an ATA assay result from at least one post-baseline sample.
Measure: Number; unit: Percentage of participants
Arm/Group | Trastuzumab Emtansine + Atezolizumab
Number analyzed (Participants) | 131
Percentage of participants | 18.3

11. Secondary Outcome: Percentage of Participants With ATAs to Trastuzumab Emtansine
Description: ATAs are antibodies that inactivate the therapeutic effects of Trastuzumab Emtansine. Patients are considered to be ATA positive if they are ATA negative at baseline but develop an ATA response following study drug administration (treatment-induced ATA response), or if they are ATA positive at baseline and the titer of one or more post-baseline samples is at least 4-fold greater (i.e., ≥ 0.60 titer units) than the titer of the baseline sample (treatment-enhanced ATA response).
Time Frame: Pre-infusion (0 h) on Day 1 Cycles 1 and 4 (each cycle = 21 days); and at any time during study treatment/early discontinuation visit (approximately 40 months)
Population: The analysis population included a patient with an ATA assay result from at least one post-baseline sample
Measure: Number; unit: Percentage of Participants
Arm/Group | Trastuzumab Emtansine + Placebo | Trastuzumab Emtansine + Atezolizumab
Number analyzed (Participants) | 60 | 129
Percentage of Participants | 0 | 2.3

ADVERSE EVENTS:
Time Frame: Baseline up to study completion, approximately 40 months
Description: The safety population is defined as all participants who received at least one dose of the study medication.
Arm/Group | Trastuzumab Emtansine + Atezolizumab | Trastuzumab Emtansine + Placebo
All-Cause Mortality (participants affected / at risk) | 42/133 | 22/67
Serious Adverse Events (participants affected / at risk) | 52/133 | 16/67
Other Adverse Events (participants affected / at risk) | 130/133 | 62/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trastuzumab Emtansine + Atezolizumab (N=133) | Trastuzumab Emtansine + Placebo (N=67)
Pneumonia (Infections and infestations) | 4 (4) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 2 (2) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 10 (12) | 0 (0)
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 1 (1) | 0 (0)
Abscess jaw (Infections and infestations) | 1 (1) | 0 (0)
Breast cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Catheter site infection (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 2 (2)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 2 (5)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (3) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Brain oedema (Nervous system disorders) | 2 (2) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1)
IgA nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trastuzumab Emtansine + Atezolizumab (N=133) | Trastuzumab Emtansine + Placebo (N=67)
Anaemia (Blood and lymphatic system disorders) | 24 (30) | 6 (7)
Neutropenia (Blood and lymphatic system disorders) | 13 (21) | 4 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 42 (105) | 12 (22)
Constipation (Gastrointestinal disorders) | 29 (38) | 10 (15)
Diarrhoea (Gastrointestinal disorders) | 34 (50) | 15 (18)
Dyspepsia (Gastrointestinal disorders) | 14 (21) | 3 (3)
Nausea (Gastrointestinal disorders) | 51 (84) | 29 (37)
Stomatitis (Gastrointestinal disorders) | 13 (21) | 2 (2)
Vomiting (Gastrointestinal disorders) | 27 (36) | 15 (19)
Nasopharyngitis (Infections and infestations) | 15 (20) | 6 (8)
Fall (Injury, poisoning and procedural complications) | 10 (14) | 3 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 26 (37) | 8 (9)
Myalgia (Musculoskeletal and connective tissue disorders) | 24 (26) | 10 (16)
Dizziness (Nervous system disorders) | 18 (18) | 9 (10)
Dysgeusia (Nervous system disorders) | 6 (6) | 5 (6)
Headache (Nervous system disorders) | 38 (62) | 17 (27)
Paraesthesia (Nervous system disorders) | 9 (16) | 2 (2)
Anxiety (Psychiatric disorders) | 2 (2) | 6 (6)
Insomnia (Psychiatric disorders) | 14 (15) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 25 (28) | 10 (12)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 (19) | 5 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 28 (39) | 10 (13)
Pruritus (Skin and subcutaneous tissue disorders) | 23 (30) | 4 (5)
Rash (Skin and subcutaneous tissue disorders) | 32 (42) | 6 (11)
Hypertension (Vascular disorders) | 4 (4) | 4 (4)
Hypothyroidism (Endocrine disorders) | 18 (19) | 3 (3)
Dry eye (Eye disorders) | 11 (12) | 4 (4)
Lacrimation increased (Eye disorders) | 7 (9) | 1 (1)
Vision blurred (Eye disorders) | 7 (8) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 17 (20) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 10 (10) | 3 (8)
Dry mouth (Gastrointestinal disorders) | 22 (23) | 9 (10)
Asthenia (General disorders) | 23 (35) | 5 (6)
Chills (General disorders) | 19 (27) | 6 (8)
Fatigue (General disorders) | 53 (87) | 30 (43)
Influenza like illness (General disorders) | 12 (16) | 8 (8)
Mucosal inflammation (General disorders) | 16 (21) | 1 (1)
Oedema peripheral (General disorders) | 7 (9) | 4 (4)
Pyrexia (General disorders) | 44 (72) | 12 (18)
Sinusitis (Infections and infestations) | 7 (9) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 18 (28) | 9 (12)
Urinary tract infection (Infections and infestations) | 9 (10) | 8 (10)
Alanine aminotransferase increased (Investigations) | 31 (44) | 13 (18)
Aspartate aminotransferase increased (Investigations) | 40 (56) | 14 (19)
Blood alkaline phosphatase increased (Investigations) | 11 (12) | 6 (8)
Gamma-glutamyltransferase increased (Investigations) | 7 (7) | 2 (2)
Weight decreased (Investigations) | 13 (13) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 30 (52) | 12 (14)
Hypokalaemia (Metabolism and nutrition disorders) | 13 (16) | 4 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 15 (19) | 8 (9)
Bone pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 3 (8)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 10 (13) | 7 (8)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 10 (12) | 6 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 (10) | 4 (5)
Neuropathy peripheral (Nervous system disorders) | 18 (20) | 7 (8)
Peripheral sensory neuropathy (Nervous system disorders) | 11 (11) | 5 (6)
Polyneuropathy (Nervous system disorders) | 2 (2) | 4 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 11 (12) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights

DOCUMENTS (2):
  • Study Protocol (2017-08-09): https://cdn.clinicaltrials.gov/large-docs/83/NCT02924883/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-16): https://cdn.clinicaltrials.gov/large-docs/83/NCT02924883/SAP_001.pdf